CLINICAL TRIAL: NCT04461769
Title: Electrical Synchronization of Slow Oscillations to Enhance Deep Sleep
Acronym: ESSOTEDS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brain Electrophysiology Laboratory Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R44MH115955 (NIH)
Record Dates: First submitted 2020-06-30; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Sleep; Sleep Hygiene
MeSH Terms: conditions — Sleep Hygiene | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: First night adaptation sleep; second and third nights (one week apart) stimulation or placebo control (order randomized).
Who Masked: Participant, Care Provider
Masking Description: Participants were blind to which night was stimulation. Experimenters were blinded until the participant was asleep, when they opened an email that specified delivery of stimulation or sham.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slow Oscillation Synchronization with TES (Experimental): Transcranial Electrical Stimulation, 0.5 Hz sine wave, 0.5 mA, between frontal (frontopolar and inferior lateral frontal) and posterior (mastoid and occipital) electrodes.
  Interventions: Device: Transcranial Electrical Stimulation
- Sham Control (Sham Comparator): No current delivered.
  Interventions: Device: Transcranial Electrical Stimulation

INTERVENTIONS:
Device: Transcranial Electrical Stimulation — Oscillating electrical current
  Other Names: Sleep WISP (Wireless Interface Sensor Pod)

SUMMARY:
This study applied slowly oscillating (0.5 hz) transcranial electrical stimulation (TES; frontopolar and lateral frontal electrodes versus mastoid and occipital electrode returns) to synchronize the endogenous slow oscillations (SOs) of deep sleep (N3 or stage 3 Non-REM). A double-blind placebo control provided no stimulation. The primary endpoint was duration of N3 sleep during the night. Thirteen normal adults completed the study (before the study was terminated because of COVID-19), and usable data were obtained from ten. The synchronizing stimulation resulted in significantly longer N3 sleep compared to placebo.

DETAILED DESCRIPTION:
Previous studies have demonstrated successful synchronization of SOs with slow TES pulses. However, the stimulation in those studies used electrodes in dorsolateral frontal areas (F3, F4 versus contralateral mastoids), consistent with the assumption that human SOs emanate from frontal neocortex. In the present study, we hypothesized that transcranial electrical stimulation (TES) could be applied to frontopolar and inferior frontal head sites in order to synchronize the limbic sources of SOs specifically and thereby enhance the duration of N3 sleep. Furthermore, based on our computational modeling with this more optimal targeting of the limbic sites, we hypothesized that we could use lower TES current levels (0.5 mA versus 1 or 2 mA in previous studies) that would be unlikely to disrupt sleep and that may still be successful in synchronizing SOs to enhance the adaptive neurophysiology of deep sleep.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* history of seizures
* epilepsy
* brain trauma or injury
* insomnia
* sleep apnea
* medications that may affect the EEG.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
N3 Duration | Measured during the night of sleep (typically 8 hours)
  Duration in minutes of N3 sleep

SECONDARY OUTCOMES:
N3 Percentage | Measured during the night of sleep (typically 8 hours)
  Percentage of the night's sleep spent in N3

CONTACTS AND LOCATIONS:
Locations (1):
- Brain Electrophysiology Laboratory Company, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No